CLINICAL TRIAL: NCT03287050
Title: FAST: Feasibility Trial of Anti-PD(L)1 and SBRT in the Treatment of Advanced, Platinum-Refractory Urothelial Carcinoma
Brief Title: Anti-PD(L)1 and SBRT in the Treatment of Advanced, Platinum-Refractory Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to changing therapeutic landscape in metastatic bladder cancer and lack of radiation/immunotherapy systemic synergy in other malignancies
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.069; HUM00135161 (Other: University of Michigan)
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab + SBRT (Experimental)
  Interventions: Drug: Pembrolizumab; Radiation: SBRT

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV q 21 days
Radiation: SBRT — Stereotactic body radiation therapy (SBRT) that will commence not later than the initiation of the second cycle of pembrolizumab. SBRT dose and fractionation will be at the discretion of the treating radiation oncologist, and will be selected to respect the normal tissue tolerance of adjacent organs at risk.

SUMMARY:
This is a feasibility trial of anti-PDL1/PD1 (pembrolizumab) and stereotactic body radiation therapy (SBRT) in patients with advanced, platinum-refractory urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologic diagnosis of urothelial carcinoma
* Subjects must have radiologic evidence of metastatic disease with measurable disease by RECIST 1.1 criteria other than the target lesion(s) for SBRT
* Subjects must have at least 1 metastatic lesion previously not radiated that is amenable to SBRT per treating radiation oncologist.
* Subjects must have had progression of disease within 12 months of platinum-containing chemotherapy (chemotherapy could have been given in the neoadjuvant, adjuvant or metastatic setting) for urothelial cancer
* ECOG performance status of 0 to 2 (Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.)
* Absolute neutrophil count of ≥ 1000/mm3, platelet count ≥ 100,000/mm3, hemoglobin ≥ 8.0 g/dl; total bilirubin/ALT/AST < 2.5 x upper limit of normal (patients with known gilbert disease who have serum bilirubin ≤3x ULN may be enrolled); serum creatinine <3.0mg/dl or if elevated, a calculated estimated glomerular filtration rate (eGFR) of ≥30 mL/min/1.73 m2
* Subjects must have recovered to baseline or ≤ grade 1 CTCAE v 4.03 from toxicities related to any prior treatments unless AE(s) are clinically non-significant and/or stable on supportive therapy
* Subjects must be ≥ 2 weeks from most recent systemic therapy or most recent radiation therapy
* Women of childbearing potential must have a negative serum or urine pregnancy test within 28 days prior to registration.
* Age ≥ 18 years

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1 and anti-CTLA-4 is NOT allowed. Prior intravesical BCG (Bacillus Calmette-Guerin) therapy is allowed
* Treatment with any investigational agent or on an interventional clinical trial within 30 days prior to registration.
* No prior or concurrent malignancy is allowed except for: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, localized or locally advanced prostate cancer definitively treated without recurrence or with biochemical recurrence only, or any other cancer fully treated or from which the subject has been disease-free for at least 2 years.
* Autoimmune diseases such as rheumatoid arthritis are NOT allowed. Vitiligo, mild psoriasis (topical therapy only) or hypothyroidism are allowed
* Need for systemic corticosteroids >10mg prednisone daily or equivalent alternative steroid
* Any history of organ allografts
* Any history of HIV or hepatitis B infection
* Known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachery Reichert, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab + SBRT
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + SBRT
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Receive 4 Doses of Pembrolizumab and at Least One Session of Treatment of SBRT
Description: Feasibility will be determined by the percentage of subjects who receive 4 doses of pembrolizumab and at least one session of treatment of SBRT (Stereotactic Body Radiation Therapy) within 15 weeks from the first dose of pembrolizumab.
Time Frame: 15 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab + SBRT
Number analyzed (Participants) | 6
percentage of participants | 83

2. Secondary Outcome: The Number of Grades 3-5 Drug Related Adverse Events (AEs)
Description: The number of grades 3-5 drug related adverse events (AEs) will be recorded. AEs will be graded using the CTCAE v4.03
Time Frame: 30 days post last dose
Measure: Number; unit: events
Arm/Group | Pembrolizumab + SBRT
Number analyzed (Participants) | 6
events | 0

3. Secondary Outcome: The Percentage of Patients That Respond to Treatment
Description: The percentage of patients that achieve either a complete response (CR) or partial response (PR). Response will be reported separately using RECIST and irRECIST criteria.
  CR (RECIST): Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions CR (irRECIST): Disappearance of all lesions in two consecutive observations not less than 4 wk apart PR (RECIST): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions PR (irRECIST): ≥50% decrease in tumor burden compared with baseline in two observations at least 4 wk apart
Time Frame: 51 weeks (up to 17, 3 week doses)
Population: One patient who did not have non-radiated measurable disease is not included.
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab + SBRT
Number analyzed (Participants) | 5
percentage of participants
  RECIST | 40
  irRECIST | 40

4. Secondary Outcome: Progression Free Survival (PFS) Time
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progressive disease (PD), or death, whichever occurs first, up to 24 months.
  PD (RECIST): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions PD (irRECIST): At least 25% increase in tumor burden compared with nadir (at any single time point) in two consecutive observations at least 4 wk apart
Time Frame: 24 months
Population: One patient who did not have non-radiated measurable disease is not included in the results table.
Measure: Number; unit: months
Arm/Group | Pembrolizumab + SBRT
Number analyzed (Participants) | 5
months
  Patient 1 | 23
  Patient 2 | 10
  Patient 3 | 2
  Patient 4 | NA — This patient was continuing treatment without progression at the time of study completion/data cut-off.
  Patient 5 | 6

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 16 month period.
Arm/Group | Pembrolizumab + SBRT
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + SBRT (N=6)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + SBRT (N=6)
Abdominal pain (Gastrointestinal disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 3
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Edema limbs (General disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hematoma (Vascular disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Infections and infestations - Other (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 2
Lymphocyte count decreased (Investigations) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Papulopustular rash (Infections and infestations) | 2
Paresthesia (Nervous system disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Personality change (Psychiatric disorders) | 1
Platelet count decreased (Investigations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash pustular (Infections and infestations) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Serum amylase increased (Investigations) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Somnolence (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Urinary urgency (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 1

LIMITATIONS AND CAVEATS:
This study was closed early (at 6 patients) due to changing therapeutic landscape in metastatic bladder cancer and lack of radiation/immunotherapy systemic synergy in other malignancies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03287050/Prot_SAP_000.pdf